CLINICAL TRIAL: NCT05759533
Title: Evaluation of the Corrected Carotid Flow Time and the Inferior Vena Cava Collapsibility Index in Predicting Post-spinal Anesthesia Hypotension in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate Professor of Anesthesiology, Fayoum University Hospital
Other Study IDs: D 316
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Corrected carotid flow time, IVC diameter — Corrected carotid flow time correction: is the carotid systole time, with heart rate correction applied IVC Collapsibility Index measurement is a reliable predictor of intraoperative hypotension within 30 minutes of spinal anesthetic administration

SUMMARY:
We include patient who will undergo elective surgeries such as orthopedic surgeries as fixator placement, lower extremity debridement, inguinal hernia, Urosurgery as bladder- prostate resection, hysterectomy, fibroid removal, ovarian cyct removal, plastic surgeries, and other types of surgery. The fasting durations of the included patients will be 8 hours for solids and 2 hours for clear liquids. There won't be any premedication given. The patient will be placed in a supine, neutral-head resting posture in the operating room as well as standard monitors such as a five-lead electrocardiography, pulse oximeter, and noninvasive blood pressure. An attending anesthesiologist will use a 25-gauge Quincke spinal needle to induce spinal anesthesia in the L3/4 or L4/5 vertebral interspace with the patient in the right lateral decubitus posture. Throughout the course of the trial, the attending anesthesiologist will choose the dosages of 0.5% hyperbaric bupivacaine (10 to 15 mg) and fentanyl (10 to 20 mg) 28. The patient will be placed back in the supine position without any lateral tilt once the spinal injection has been given over a period of 15 to 30 seconds. Three minutes following the spinal injection, the sensory block will be evaluated with a cold and pinprick test. The mean blood pressure will be taken every 3 minutes between the spinal injection and delivery, and every 5 minutes from the delivery until the end of the procedure. The lowest SBP measured between the spinal anesthesia injection and delivery will be determined, together with the percentage of the SBP drop from the pre-anesthetic SBP. The patient's head will be turned 308 degrees to the left. First, a 6.0 to 13.0MHz linear array transducer will be positioned vertically on the neck with the probe marker facing the patient's head. The lower edge of the thyroid cartilage will provide a long-axis B-mode picture of the right common carotid artery. The probe will then be positioned in the lumen's center, around 2 cm from where the carotid arteries split. After that, carotid artery blood flow waveforms will be preserved together with a pulsed Wave-Doppler trace of the artery's flow. The cycle time will be determined by counting the number of heartbeats at the start of the systolic upstroke using an ultrasound machine's caliper function. By taking measurements in one-tenth of millisecond intervals between the systolic upstroke and the diastolic notch, the flow time will be determined. the IVC will be scanned using a portable ultrasound device (LOGIQ-e by GE health care) and a 3.5-5 MHz curvilinear probe in the subxiphoid region (paramedian long-axis view), just close to the common hepatic vein's draining to the IVC. At the point where the IVC joins the right atrium, a 2D picture will be obtained. M-mode imaging will be used to record changes in IVC diameter during inspiration and expiration. The procedure is carried out two to three centimeters away from the right atrium/IVC junction. The attending anesthetist will keep track of how long it took to locate the IVC after placing the probe on the patient. The M mode of the ultrasonography will be used to measure the IVC's Minimum (IVCDMin) and Maximum (IVCDMax) diameters, and the IVC Collapsibility Index (IVCCI) will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients age above 60 years old.
* Patients had no contraindications for spinal anesthesia.
* Patients undergoing elective surgery.

Exclusion Criteria:

* Patients with a BMI of more than 35 Kg/m2.
* Patients suffering from carotid stenosis.
* Patients with systolic blood pressure greater than 160 mmHg.
* Patients who need preoperative hydration.
* Patients undergoing emergency surgery

Ages: 60 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Geriatric patients during elective surgeries.
Sampling Method: Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
ROC under the curve | From 1 December, 2022 to 1 December, 2023
  Receiver operating characteristic (ROC) under the curve with the best cut-off of the value of the corrected carotid flow time and IVC collapsibility index in predicting PSAH in geriatric patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No